CLINICAL TRIAL: NCT03484117
Title: Addressing Barriers to Retention in HIV Care for Hispanic Immigrants
Brief Title: Retention in HIV Care for Hispanic Immigrants
Acronym: ADELANTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Julie H Levison, MD, MPhil, MPH, Assistant Professor of Medicine at Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016P000252; 5K23MH100978-04 (NIH)
Record Dates: First submitted 2018-03-07; First posted 2018-03-30 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Community Health Workers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention): Participants in this arm will receive bilingual written materials on healthy living with HIV at the baseline visit. At baseline and exit, all participants will be assessed using instruments to measure demographics and self-perceived barriers to care for Hispanic immigrants.
- Community Health Worker (Experimental): Participants in the intervention arm will receive 5 one-on-one sessions over 24 weeks with a Spanish-speaking CHW. At baseline and exit, all participants will be assessed using instruments to measure demographics and self-perceived barriers to care for Hispanic immigrants
  Interventions: Behavioral: Community Health Worker

INTERVENTIONS:
Behavioral: Community Health Worker — Participants will receive 5 one-on-one sessions with a CHW over 24 weeks.
  Arms: Community Health Worker

SUMMARY:
A randomized trial to test the feasibility and acceptability of an intervention to improve retention in HIV primary care in HIV-infected Hispanic immigrants compared to a "treatment as usual" condition. We will measure feasibility, acceptability, study retention, and effect sizes of outcomes in order to inform a larger trial. The intervention design is based on qualitative research with HIV-infected Hispanic immigrants and their HIV providers. The intervention will be led by a Spanish-speaking community health worker trained in HIV health promotion.

DETAILED DESCRIPTION:
Overview:

Participants will be HIV-infected Hispanic immigrants age ≥18 years. Participants will be recruited from Partners-affiliated infectious disease and primary care clinics as well as clinics and community-based organizations in the Greater Boston area with high contact with HIV-infected Hispanics. In the intervention, a bilingual (English-Spanish speaking) community health worker (CHW) will deliver personalized sessions framed around a Spanish-language multi-media health communication tool. The CHW will deliver the intervention over a 16 to 24 week period.

Study procedures:

Participants will be HIV-infected Hispanic immigrants age ≥18 years at risk for inconsistent attendance (as measured during study screening). Participants will be recruited via provider referral, peer referral, flyers, and social media. Once an individual expresses interest in the study, a study staff member will screen that individual to assess eligibility. Individuals who are eligible will be invited to enroll through an informed consent process and complete a baseline survey. After completion of the baseline survey, study staff will randomize participants into a treatment as usual (TAU) group or intervention group. At trial exit, all participants, including the TAU group, will complete an in-depth assessment to measure their barriers to HIV care and provide feedback about their experience in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older and able to communicate in Spanish or English
* Born in Puerto Rico or Spanish-speaking Latin American country
* HIV-infected or HIV-positive
* New HIV diagnosis or unable to regularly attend HIV primary care appointments

Exclusion Criteria:

* Unable to provide verbal consent due to unstable medical or psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie H Levison, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment as Usual | Community Health Worker
Started | 32 | 35
Completed | 30 | 31
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 1 | 3
Not completed — Declined participation in exit assess | 1 | 1

BASELINE CHARACTERISTICS:
Population: Data obtained from 67 participants who enrolled and completed baseline assessment
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual | Community Health Worker | Total
Number analyzed (Participants) | 32 | 35 | 67
Age, Customized [Count of Participants; unit: Participants]
  18-25 years | 1 | 3 | 4
  >=26 years | 31 | 32 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 28
  Male | 22 | 17 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 35 | 67
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 5 | 3 | 8
  More than one race | 19 | 22 | 41
  Unknown or Not Reported | 4 | 6 | 10
HIV Viral suppression [Count of Participants; unit: Participants] — Number of participants with HIV RNA <200 copies/ml Population: Number of individuals analyzed were the total number of participants with available laboratory data.
  Participants
    number analyzed (Participants) | 31 | 35 | 66
    (all) | 27 | 31 | 58
Baseline CD4 cell count [Count of Participants; unit: Participants] — Population: Number of participants analyzed were the total number of participants with available laboratory data.
  Participants
    number analyzed (Participants) | 31 | 35 | 66
    0-200 cells/mm^3 | 1 | 3 | 4
    201-500 cells/mm^3 | 11 | 7 | 18
    >500 cells/mm^3 | 19 | 25 | 44

OUTCOME MEASURES:

1. Primary Outcome: Retention in Care - Yes Responses
Description: A dichotomized outcome (yes/no) with yes defined as at least one visit to HIV clinic at both time periods (week 1-16 and week 17-32), and no defined as no HIV visit from at least one time period. Responses determined by review of the medical record for evidence of attended HIV clinic visits.
Time Frame: 32 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual | Community Health Worker
Number analyzed (Participants) | 32 | 35
Participants | 19 | 23

2. Secondary Outcome: Number of Participants With HIV Viral Load Suppression up to Week-24
Description: Participants with HIV viral load <200 copies/ml
Time Frame: From baseline to week-24
Population: HIV viral load laboratory data at week-24 available for a total of 66 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual | Community Health Worker
Number analyzed (Participants) | 31 | 35
Participants | 30 | 31

3. Secondary Outcome: Change in CD4 T-cell Count Over 24 Weeks
Description: Change in CD4 T-cell count from baseline to week-24 post-randomization
Time Frame: From baseline to week-24
Population: CD4 count laboratory data at week-24 available for 66 participants.
Measure: Mean (Standard Deviation); unit: 1000 cells/uL
Arm/Group | Treatment as Usual | Community Health Worker
Number analyzed (Participants) | 31 | 35
1000 cells/uL | 6.0 (174.8) | 25.7 (137.0)

4. Secondary Outcome: Number of Participants With HIV Viral Load Suppression up to 48 Weeks.
Description: Number of participants with HIV RNA <200 copies/ml
Time Frame: Baseline to week-48
Population: HIV viral load laboratory data at week-48 available for 59 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual | Community Health Worker
Number analyzed (Participants) | 28 | 31
Participants | 27 | 26

5. Secondary Outcome: Change in CD4 T-cell Count Over 48 Weeks.
Description: Change in CD4 T-cell count from baseline to week-48 post-randomization
Time Frame: Baseline to week-48
Population: CD4 count laboratory data at week-48 available for 59 participants.
Measure: Mean (Standard Deviation); unit: 1000 cells/uL
Arm/Group | Treatment as Usual | Community Health Worker
Number analyzed (Participants) | 28 | 31
1000 cells/uL | -2.4 (179.4) | 29.6 (184.6)

ADVERSE EVENTS:
Time Frame: through study completion up to 48 weeks
Arm/Group | Treatment as Usual | Community Health Worker
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/35
Other Adverse Events (participants affected / at risk) | 0/32 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT03484117/Prot_SAP_000.pdf